CLINICAL TRIAL: NCT02003495
Title: Immunogenicity and Safety of Meningococcal (A, C, Y and W135) Conjugate Vaccine in Healthy Subjects 2 Months to 6 Years of Age in China
Brief Title: Immunogenicity and Safety of Meningococcal (A, C, Y and W135) Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013L01041; 2013L01041 (Registry Identifier: China food and drug administration)
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Meningitis
Keywords: Immunogenicity, Safety, Meningococcal Conjugate Vaccine
MeSH Terms: conditions — Meningitis | interventions — Vaccines, Conjugate; serogroup C meningococcal conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- MCV-ACYW135 Vaccine Group (Experimental): Participants at age 2 to 6 years of enrollment will receive 1 dose on Meningococcal ( A, C, Y and W 135) conjugate vaccine.
  Participants at age 6 to 23 months of enrollment will receive 2 doses on Meningococcal ( A, C, Y and W 135) conjugate vaccine at 3 months apart.
  Participants at age 3 to 5 months of enrollment will receive 3 doses on Meningococcal ( A, C, Y and W 135) conjugate vaccine at 1 month apart.
  Participants at age 2 to 5 months of enrollment will receive 3 doses on Meningococcal ( A, C, Y and W 135) conjugate vaccine at 2 months apart.
  Interventions: Biological: MCV-ACYW135 Vaccine Group
- MPV-ACYW135 Vaccine Group (Active Comparator): Participants at age 2 to 6 years of enrollment will receive 1 dose on Group A, C, Y and W135 Meningococcal Polysaccharide Vaccine
  Interventions: Biological: MPV-ACYW135 Vaccine Group
- MPV-A Vaccine Group (Active Comparator): Participants at age 6 to 23 months of enrollment will receive 2 doses on Group A Meningococcal Polysaccharide vaccine at 3 months apart.
  Interventions: Biological: MPV-A Vaccine Group
- MCV-AC Vaccine Group (Active Comparator): Participants at age 3 to 5 months of enrollment will receive 3 doses on Group A and C Meningococcal conjugate vaccine at 1 month apart.
  Interventions: Biological: MCV-AC Vaccine Group
- Hib Vaccine Group (Placebo Comparator): Participants at age 2 to 5 months of enrollment will receive 3 doses on Haemophilus Influenzae Type b Conjugate Vaccine at 2 months apart.
  Interventions: Biological: Hib Vaccine Group

INTERVENTIONS:
Biological: MCV-ACYW135 Vaccine Group — 0.5ml, intramuscular
  Other Names: Meningococcal ( A, C, Y and W 135) conjugate vaccine
  Arms: MCV-ACYW135 Vaccine Group
Biological: MPV-ACYW135 Vaccine Group — 0.5ml, intramuscular
  Other Names: Group A, C, Y and W-135 Meningococcal Polysaccharide Vaccine
  Arms: MPV-ACYW135 Vaccine Group
Biological: MPV-A Vaccine Group — 0.5ml, intramuscular
  Other Names: Group A Meningococcal Polysaccharide vaccine
  Arms: MPV-A Vaccine Group
Biological: MCV-AC Vaccine Group — 0.5ml, intramuscular
  Other Names: Group A and C Meningococcal conjugate vaccine
  Arms: MCV-AC Vaccine Group
Biological: Hib Vaccine Group — 0.5ml, intramuscular
  Other Names: Haemophilus Influenzae Type b Conjugate Vaccine
  Arms: Hib Vaccine Group

SUMMARY:
The purpose of this observer-blind study is to evaluate the safety, reactogenicity and immunogenicity of Meninggococcal (A,C,Y and W135) Conjugate Vaccine in 2 months to 6 years-old children.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol should be enrolled in the study.
* Healthy permanent residence 2 months to 6 years old.
* Subjects and parent/guardian able to attend all scheduled visits and comply with all study procedures.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* History of meningitis infection or vaccination of meningococcal vaccine within the past 6 months.
* Allergic history or any SAE after vaccination, such as allergy, urticaria, dyspnea, angioedema, celialgia.
* Patients administered with immunosuppressive agents, cytotoxicity factor or corticosteroids in the 6 months preceding the vaccine trial.
* Receipt of blood or blood-derived products in the 3 months preceding vaccination
* Participation in another clinical study investigating a vaccine, drug in the 30 days preceding vaccination.
* Receipt of any live virus vaccine in the 15 days preceding vaccination.
* Receipt of any subunit vaccine and inactivated vaccine in the 7 days before vaccination.
* Febrile illness (temperature ≥ 38°C) in the 3 days or any acute illness/infection in the 7 days preceding vaccination.
* Thrombocytopenia.
* History of thyroid gland excision or treatment for thyroid gland disease in last 12 months.
* Functional or anatomic asplenia.
* History of eclampsia, epilepsy, encephalopathy and mental disease or family disease.
* Chronic disease (such as Down syndrome, diabetes, sickle cell anemia or neurologic disease, Guillain-Barre Syndrome).
* Known or suspected diseases, including: respiratory system disease, acute infection or active stage of chronic disease, HIV infection of children or mothers, cardiovascular disease, acute hypertension, cancer treatment, skin disease, etc.
* Any condition that, in the judgment of investigator, may affect trial assessment.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2195 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects exhibiting a >= 4fold increase in rSBA titers level from pre-vaccination to post-vaccination | 28 days after vaccination

SECONDARY OUTCOMES:
to evaluate the adverse reactions after vaccination | Within 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: shengli xia, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Zhengzhou, Henan, China